CLINICAL TRIAL: NCT00293683
Title: Cesarean Delivery Skin Closure: A Randomized Controlled Trial of Standard Staples Versus Absorbable Staples
Brief Title: A Study Comparing Two Different Techniques for Closing the Skin After a Cesarean Delivery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Thomas Jefferson University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 04U.498
Record Dates: First submitted 2006-02-16; First posted 2006-02-17 (Estimated); Last update posted 2014-07-29 (Estimated); Status verified 2014-07

CONDITIONS: Cesarean Section
Keywords: cesarean; closure; skin; staple; absorbable; metal

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: Insorb absorbable skin staple

SUMMARY:
We hypothesize that the use of absorbable staples to close cesarean skin incisions will cause less pain, have better long-term cosmetic results, and result in improved patient satisfaction over standard metal staples. We expect to see no difference in wound complication rates with these two cesarean skin closure techniques.

DETAILED DESCRIPTION:
Type: Randomized controlled trial

Selection of Patients: All pregnant women, undergoing a primary (their first) cesarean delivery at Thomas Jefferson University Hospital will be offered randomization regardless of indication for cesarean delivery. Patients will be excluded from the study if they have a history of a previous cesarean delivery, history of a previous Pfannensteil skin incision for an indication other than for a cesarean delivery (i.e. myomectomy, laparotomy), or a planned vertical skin incision prior to randomization.

Randomization:

Patients will be randomized to skin closure with either the standard staples or the Insorb™ absorbable staple using a computer-generated random number sequence in blocks of six and ten. Allocation will be concealed in opaque, sealed study envelopes that are held on labor and delivery until after consent is obtained. Patients will not be masked as to the type of stapler used however, the investigator obtaining outcome data at six months will be masked.

Procedure:

The cesarean delivery should be performed in the usual fashion according to the surgeon's preference.

We recommend:

* Skin is prepped with a suitable antibacterial agent
* Appropriate prophylactic antibiotics
* Bladder flap should not be routinely created or closed
* Uterus may be closed in 1 or 2 layers
* Peritoneum should not be routinely closed
* Skin wound should be irrigated after fascia closure
* Subcutaneous drains or sutures at surgeon's discretion
* Steri-strips will be placed prior to dressing placement in the OR
* Dressing removal on POD #1
* Metal staple removal prior to discharge from hospital preferred, but ultimately up to surgeon's discretion

Skin incisions will be closed with the assigned stapling device. Addison tissue forceps will be used to evert the skin edges. The recommended distance between staples is 8 to 10mm; however this can be altered at the discretion of the operating physician.

Follow Up:

The subject's age, race, gravidity, parity, reported weight, indication for cesarean delivery, medical co-morbidity, delivery associated complications and findings, charted pain medication and clinic status will be assessed by chart review. Pain, time of placement, patient satisfaction, and cosmetic outcome will be assessed by data sheets filled out by the OR staff, physicians, and patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients at TJUH undergoing primary cesarean delivery via Pfannenstiel incision
* Surgeon willing to adhere to randomized skin staple category

Exclusion Criteria:

* Known allergy to staples or suture
* Vertical skin incision
* Repeat cesarean deliveries

Ages: 12 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 120
Dates: Start 2004-12; Primary Completion 2014-10 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Post operative pain

SECONDARY OUTCOMES:
Length of time of skin closure
Costs
Cosmetic outcome
Wound disruption rate
Infection rate
Patient Satisfaction

CONTACTS AND LOCATIONS:
Overall Officials: Jason K. Baxter, MD, MSCP, Principal Investigator — Thomas Jefferson University
Locations (1):
- Thomas Jefferson University Hospital, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Background] Frishman GN, Schwartz T, Hogan JW. Closure of Pfannenstiel skin incisions. Staples vs. subcuticular suture. J Reprod Med. 1997 Oct;42(10):627-30. PMID 9350017
- [Background] Ranaboldo CJ, Rowe-Jones DC. Closure of laparotomy wounds: skin staples versus sutures. Br J Surg. 1992 Nov;79(11):1172-3. doi: 10.1002/bjs.1800791122. PMID 1467895
- [Background] Alderdice F, McKenna D, Dornan J. Techniques and materials for skin closure in caesarean section. Cochrane Database Syst Rev. 2003;(2):CD003577. doi: 10.1002/14651858.CD003577. PMID 12804476
- [Background] Fick JL, Novo RE, Kirchhof N. Comparison of gross and histologic tissue responses of skin incisions closed by use of absorbable subcuticular staples, cutaneous metal staples, and polyglactin 910 suture in pigs. Am J Vet Res. 2005 Nov;66(11):1975-84. doi: 10.2460/ajvr.2005.66.1975. PMID 16334959
- [Background] Pickford IR, Brennan SS, Evans M, Pollock AV. Two methods of skin closure in abdominal operations: a controlled clinical trial. Br J Surg. 1983 Apr;70(4):226-8. doi: 10.1002/bjs.1800700414. PMID 6338996
- [Background] Zwart HJ, de Ruiter P. Subcuticular, continuous and mechanical skin closure: cosmetic results of a prospective randomized trial. Neth J Surg. 1989 Jun;41(3):57-60. No abstract available. PMID 2501713